CLINICAL TRIAL: NCT07074990
Title: Clinical Study Evaluating the Efficacy and Safety of Colchicine in Adult Patients With Sepsis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Randa Hamza Ismail Elmohr, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: colchicine in sepsis
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Sepsis at Intensive Care Unit
Keywords: Sepsis, Inflammation, Colchicine, Serum Tumor necrosis factor-alpha (TNF-α),Serum Malondialdehyde (MDA),Sequential Organ Failure Assessment (SOFA) score
MeSH Terms: conditions — Sepsis; Inflammation | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, and controlled parallel design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Control group) (Placebo Comparator)
  Interventions: Drug: conventional sepsis therapy alone
- Group 2 (Colchicine group) (Active Comparator)
  Interventions: Drug: colchicine 500 mcg oral twice daily plus conventional sepsis therapy.

INTERVENTIONS:
Drug: conventional sepsis therapy alone — fluid resuscitation a minimum of 30 mL/kg of intravenous (IV) crystalloid fluid administered during the initial 3 hours of resuscitation, along with empiric antibiotic therapy aimed at the suspected pathogens and infection sites, ideally starting within the first hour.
  Arms: Group 1 (Control group)
Drug: colchicine 500 mcg oral twice daily plus conventional sepsis therapy. — colchicine 500 mcg oral twice daily plus conventional sepsis therapy for 5 days.
  Arms: Group 2 (Colchicine group)

SUMMARY:
Inflammatory markers are found to be an important contributor in sepsis. We evaluate the effect of colchicine on inflammatory processes and its possible protective effect against oxidative stress and organ dysfunction in adult patients suffering from sepsis.

DETAILED DESCRIPTION:
Sepsis is life-threatening organ dysfunction caused by a dysregulated host response to infection. Sepsis and septic shock are major healthcare problems, impacting millions of people around the world each year and killing between one in three and one in six of those it affects. Early identification and appropriate management in the initial hours after the development of sepsis improve outcomes .

Large quantities of proinflammatory cytokines released in patients with sepsis may spill into the bloodstream, contributing to the progression of a local infection to sepsis. These include tumor necrosis factor alpha (TNF-α), interleukin-1 (IL-1) and, interleukin-6 (IL-6), all of them can cause fever, hypotension, leukocytosis, induction of other proinflammatory cytokines, and the simultaneous activation of coagulation and fibrinolysis.

Taken together of all the aspects of the pathogenesis of sepsis, treatment modalities with anti-inflammatory effects could be considered for the successful treatment of sepsis. The available treatment strategies for management of sepsis include the use of fluid resuscitation and Empiric antibiotic therapy .

However, the limited success of antimicrobial in reducing the high mortality associated with sepsis and septic shock, increasing antibiotic resistance and medicine-resistant hemodynamic changes and our improved understandings of the pathogenesis of sepsis have resulted in further research on new treatment modalities in addition to classical treatments .

In particular, the identification of endotoxin-induced TNF-α and IL-1 production during sepsis as a major mediator of host damage, which culminates in potentially irreversible multi-organ dysfunction and shock, has led to the experimental use of a variety of interventions .

In this condition, novel agents must be developed or old drugs could be re-purposed to provide greater therapeutic outcome with fewer side effects at a minimum cost. Considering these facts, compounds from natural products may be considered as a promising and fruitful strategy for the treatment of sepsis.

Colchicine is a tricyclic, lipid-soluble alkaloid extracted from the plant of the Lily family Colchicum autumnale. The therapeutic use of colchicine has been well documented in gout and familial Mediterranean fever. it has also been used in other diseases including Behcet's disease, pericarditis, coronary artery disease and other inflammatory and fibrotic conditions .

Hypothesis: In this context, the outcomes of the previous animal studies and pilot study can provide a proof of concept for the implication of colchicine in clinical settings in order to improve the outcome in patients with sepsis and its efficacy in management of sepsis may depend on its anti-inflammatory and antioxidant effects.

ELIGIBILITY:
* Inclusion criteria:

  * Adult age ≥18 years old.
  * Both male and female sex.
  * Patients diagnosed with sepsis regardless its etiology according to the definitions of SSC .
* Exclusion criteria:

  * Late septic shock at presentation with multiple organ failure.
  * Serious gastrointestinal disease.
  * Preexisting end stage liver disease.
  * Preexisting end stage renal disease
  * Pregnancy and breast-feeding women.
  * History of allergy or intolerance to Colchicine.
  * Patient with malignancies.
  * Uncontrolled hemorrhage.
  * Burn.
  * Patients on immunosuppressant or biological therapies.
  * Concomitant use of P-glycoprotein (P-gp) inhibitor such as: Verapamil, and Amiodarone or strong CYP3A4 inhibitor such as: Clarithromycin, Ritonavir and Ketoconazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
change in the measured biological marker Serum Tumor necrosis factor-alpha (TNF-α) . | 10 Months
  decrease in (TNF-α) level means improvement from sepsis and better outcome
change in the measured biological marker Serum Malondialdehyde (MDA). | 10 Months
  decrease in Serum Malondialdehyde (MDA) level means improvement from sepsis and better outcome.

SECONDARY OUTCOMES:
change in Sequential Organ Failure Assessment (SOFA) score | 10 Months
  decrease in Sequential Organ Failure Assessment (SOFA) score means improvement of organ dysfunction and improvement in sepsis ( better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy - Tanta University, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
scientific paper